CLINICAL TRIAL: NCT04468971
Title: Phase 1 Double-Blinded, Randomized, Placebo Controlled Safety and Early Efficacy Trial of Cryopreserved Cord Blood Derived T-Regulatory Cell Infusions (CK0802) In The Treatment Of COVID-19 Induced Acute Respiratory Distress Syndrome (ARDS)
Brief Title: REgulatory T Cell infuSion fOr Lung Injury Due to COVID-19 PnEumonia
Acronym: RESOLVE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cellenkos, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CK0802.501.1
Record Dates: First submitted 2020-07-10; First posted 2020-07-13 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: COVID19; ARDS
Keywords: COVID19; ARDS; CK0802; T regulatory cells; cord blood
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Multi-center, prospective, double-blinded, placebo controlled Phase 1 randomized clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Placebo Comparator): Excipient
  Interventions: Drug: Placebo
- Arm 2 (Experimental): CK0802: 1x10^8 cells
  Interventions: Biological: CK0802
- Arm 3 (Experimental): CK0802: 3x10^8 cells
  Interventions: Biological: CK0802

INTERVENTIONS:
Biological: CK0802 — Cryopreserved, off the shelf, cord blood derived T regulatory cells
  Arms: Arm 2; Arm 3
Drug: Placebo — Expicient
  Arms: Arm 1

SUMMARY:
To assess the safety and efficacy of CK0802 in treatment of patients with COVID-19 induced moderate-to-severe PNA-ARDS.

ELIGIBILITY:
Inclusion Criteria:

* Documented to have an RT-PCR-based diagnosis of SARS-CoV-2 infection by RT-PCR
* Moderate-to-severe ARDS as defined by the Berlin Criteria: ratio of partial pressure of arterial oxygen (PaO2) to the fraction of inspired oxygen (FiO2) of 200 mm Hg or less assessed with a positive end-expiratory pressure (PEEP) of >5 cm H2O.
* Intubated for less than 120 hours
* Age ≥18 years
* Ability to provide informed consent or duly appointment health care proxy with the authority to provide informed consent.

Exclusion Criteria:

1. In the opinion of the investigator, unlikely to survive for >48 hours from screening.
2. Any physical examination findings and/or history of any illness that, in the opinion of the study investigator, might confound the results of the study or pose an additional risk to the patient by their participation in the study.
3. Currently receiving extracorporeal membrane oxygenation (ECMO) or high frequency oscillatory ventilation (HFOV).
4. Females who are pregnant.
5. Patients with active bacteremia at start of therapy enrollment or concurrently active moderate to severe other infectious which in the opinion of the investigator may possibly affect the safety of CK0802 treatment.
6. Patients who have been intubated for more than 120 hours.
7. Known hypersensitivity to DMSO or to porcine or bovine protein.
8. Any end-stage organ disease which in the opinion of the investigator may possibly affect the safety of CK0802 treatment.
9. High dose steroids.
10. Receiving an investigational cellular therapy agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
Regimen related ≥ grade 3 toxicity within 48 hours of first infusion | 48 hours
  Regimen related ≥ grade 3 toxicity within 48 hours of first infusion (DLT)
28-day treatment success, defined as S28 | 28 days
  Alive and not intubated 28 days after the date of first infusion

SECONDARY OUTCOMES:
Time to extubation | 28 days
  Time to extubation
Oxygenation improvement | 11 days
  Oxygenation requirement (PaO2/FiO2) change between day 0 and day +11
Ventilator free days | 28 days
  Ventilator free days measured at day 28
Organ failure free days | 28 days
  Organ failure free days measured at day 28
ICU free days | 28 days
  ICU free days measured at day 28
All-cause mortality | 28 days
  All-cause mortality at day 28

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Columbia University, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Baylor College of Medicine, St Luke's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No